CLINICAL TRIAL: NCT06901050
Title: Effect of FAST HUGS WITH ICU Approach on Length of Intensive Care Unit Stay in Patients With Hypoxic Respiratory Failure: A Randomized Controlled Trial
Brief Title: Effect of FAST HUGS WITH ICU Approach on Length of Intensive Care Unit Stay in Patients With Hypoxic Respiratory Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: MuşAlparslan
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hypoxic Respiratory Failure
Keywords: Hypoxic respiratory failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The FAST HUGS WITH ICU approach will be applied to the experimental group. We plan to follow up patients with Hypoxic Respiratory Failure using the abbreviation FAST HUGS WITH ICU (Feeding, Analgesia, Sedation, Thromboembolic prophylaxis, Head of bed elevation, Stress Ulcer prophylaxis and Glucose control Spontaneous breathing trial, Water Balance and constipation, Investigation and results, Therapy, Hypo-hyper delirium, Invasive devices, Check the daily infection parameters, Use a checlist).
  Interventions: Other: FAST HUGS WITH ICU approach
- Control Group (No Intervention): The standard procedure will be applied to the control group.

INTERVENTIONS:
Other: FAST HUGS WITH ICU approach — FAST HUGS WITH ICU; It is an abbreviation of "Feeding, Analgesia, Sedation, Thromboembolic prophylaxis, Head of bed elevation, Stress Ulcer prophylaxis and Glucose control Spontaneous breathing trial, Water Balance and constipation, Investigation and results, Therapy, Hypo-hyper delirium, Invasive devices, Check the daily infection parameters, Use a checlist". With this approach, patients will be followed up.
  Arms: Experimental Group

SUMMARY:
This study will investigate the effect of the FAST HUGS WITH ICU approach on the length of stay in the intensive care unit in patients with hypoxic respiratory failure. Patients will be randomly assigned to the experimental and control groups. The standard procedure will be applied to the control group. The FAST HUGS WITH ICU approach will be applied to the experimental group. We plan to follow up patients with Hypoxic Respiratory Failure using the abbreviation FAST HUGS WITH ICU (Feeding, Analgesia, Sedation, Thromboembolic prophylaxis, Head of bed elevation, Stress Ulcer prophylaxis and Glucose control Spontaneous breathing trial, Water Balance and constipation, Investigation and results, Therapy, Hypo-hyper delirium, Invasive devices, Check the daily infection parameters, Use a checlist). The two groups will be examined in terms of hospital stay and some blood gas parameters.

DETAILED DESCRIPTION:
Hypoxic respiratory failure is responsible for 1.9 million patient admissions per year in the United States alone, and the hospital mortality rate is as high as 20%. This rate is also increasing in Turkey. The most common causes include pneumonia, cardiogenic pulmonary edema, ARDS, and chronic obstructive pulmonary disease (COPD). Fast hugs is important in affecting the prognosis of patients with hypoxic respiratory failure in special clinics such as the Chest Diseases Intensive Care Unit. Therefore, new studies are needed. This study will investigate the effect of the FAST HUGS WITH ICU approach on the length of stay in the intensive care unit in patients with hypoxic respiratory failure. Patients will be randomly assigned to the experimental and control groups. The standard procedure will be applied to the control group. The FAST HUGS WITH ICU approach will be applied to the experimental group. We plan to follow up patients with Hypoxic Respiratory Failure using the abbreviation FAST HUGS WITH ICU (Feeding, Analgesia, Sedation, Thromboembolic prophylaxis, Head of bed elevation, Stress Ulcer prophylaxis and Glucose control Spontaneous breathing trial, Water Balance and constipation, Investigation and results, Therapy, Hypo-hyper delirium, Invasive devices, Check the daily infection parameters, Use a checlist). The two groups will be examined in terms of hospital stay and some blood gas parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being in the Chest Intensive Care Unit
* Having Hypoxic Respiratory Failure

Exclusion Criteria:

* Death during hospitalization

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
length of hospital stay | 1 month
  The difference between the duration of participants' admission to the intensive care unit and the time they are discharged from the intensive care unit will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Güzel Nur YILDIZ, Dr, Study Director — Muş Alparslan University
Locations (1):
- Ataturk University Research Hospital, Erzurum, Turkey (Türkiye)